CLINICAL TRIAL: NCT02109536
Title: The Use of Magnetic Endoscopic Imagers During Colonoscopy for Loop Recognition and Resolution
Status: Terminated | Type: Observational
Why Stopped: As the study progressed, the intervention became more of a standard of care, thus the study has stalled and been aborted.
Sponsor: Lawrence Charles Hookey (Other)
Responsible Party: Sponsor-Investigator, Lawrence Charles Hookey, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Other Study IDs: DMED-1639-13
Record Dates: First submitted 2014-02-24; First posted 2014-04-10 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Colonoscopic Surgical Procedures
Keywords: Colonoscopy; Looping; Loop recognition; magnetic endoscopic imager

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Staff Gastroenterologists.: Staff Gastroenterologists ability to recognize loops will be assessed using an magnetic endoscopic imager.
  Interventions: Device: Magnetic endoscopic imager.

INTERVENTIONS:
Device: Magnetic endoscopic imager. — recognizing loop type accuracy of loop type detection methods of loop reduction assessed by type

SUMMARY:
The purpose of this study is threefold. First, the ability of experienced colonoscopists to recognize the type of loop formed will be assessed and whether the use of the MEI improves this accuracy. Second, to determine which maneuvers are used for loop reduction and whether certain loops have set ways to reduce them. The third component will assess whether the colonoscopist thought that the imager helped or not.

ELIGIBILITY:
Inclusion Criteria:

* adults (18 years and older) undergoing colonoscopy

Exclusion Criteria:

* age less than 18 years old
* not willing to participate
* cardiac pacemaker
* internal cardiac defibrillator
* previous colonic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive male and female patients, 18 years or older, undergoing outpatient colonoscopy in the MEI room at Hotel Dieu Hospital in Kingston, Ontario, Canada will be considered for the study.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-12-08 (Actual); Study Completion 2018-12-08 (Actual)

PRIMARY OUTCOMES:
Accuracy of loop recognition by experienced colonoscopists compared to the magnetic imager. | within 3 mths
  When an endoscopist encounters looping they will verbalize what type of loop they think they have and this will be recorded by the endoscopy nurse on a pre-printed data collection sheet. The magnetic imager will then be turned on and a photo of the imager loop will be saved. A physician not involved with the colonoscopy will compare the image to the endoscopist's answer to determine whether they were correct or incorrect.

SECONDARY OUTCOMES:
Qualitative description of maneuvers used for loop reduction. | within 3 mths
  When an endoscopist encounters looping they will verbalize what type of loop they think they have and what maneuvers (example, reducing with clockwise torque) they used to reduce the loop. The magnetic imager will be turned on and the endoscopist will comment on whether the imager was helpful in reducing the loop. This information will be collected on a pre-printed data collection sheet.

CONTACTS AND LOCATIONS:
Overall Officials: Aman V Arya, MD, Principal Investigator — Queen's University, GIDRU; Lawrence Hookey, MD, Principal Investigator — Queen's University, GIDRU; Stephen Vanner, MD, Principal Investigator — Queen's University, GIDRU
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada